CLINICAL TRIAL: NCT04333680
Title: Transducer Selection in the Speed and Quality of Image Acquisition in FAST Exams
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sherwin Soltani, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: H-46446
Record Dates: First submitted 2020-03-11; First posted 2020-04-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Diagnostic Abdominal Ultrasonography; Trauma Injury
Keywords: ultrasonography; FAST exam; Focused assessment of sonography for trauma; Transducer selection
MeSH Terms: conditions — Accidental Injuries | interventions — Focused Assessment with Sonography for Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Phased Array (Active Comparator): Operators who will be using a phased array-type transducer to perform the FAST exam on a healthy normal volunteer.
  Interventions: Diagnostic Test: Focused Assessment of Sonography for Trauma Exam
- Curvilinear (Active Comparator): Operators who will be using a curvilinear array-type transducer to perform the FAST exam on a healthy normal volunteer.
  Interventions: Diagnostic Test: Focused Assessment of Sonography for Trauma Exam

INTERVENTIONS:
Diagnostic Test: Focused Assessment of Sonography for Trauma Exam — Speed and image quality of ultrasound exams performed with either transducer specified in the arms.
  Other Names: FAST exam; Abdominal sonography; Abdominal ultrasonography

SUMMARY:
The Focused Assessment of Sonography for Trauma (FAST) is a rapid point-of-care ultrasound exam performed on blunt and penetrating trauma patients who are too critically injured to be transported to a CT scanner. Low-frequency ultrasound is used to image the abdomen and pericardium in these patients, using either a curvilinear transducer or a phased-array transducer. Whether the use of one transducer or the other is better for this application is not well studied. In this study, physician ultrasound operators will perform the FAST exam on healthy non-injured volunteers to determine if the speed or quality of images between the two transducer types is different.

DETAILED DESCRIPTION:
The Focused Assessment of Sonography for Trauma (FAST) is a rapid point-of-care ultrasound exam performed on blunt and penetrating trauma patients who are too critically injured to be transported to a CT scanner. In performing this exam, time to acquisition of adequate images is crucial to clinical decision-making as patients undergoing this exam have a high probability of deteriorating if not intervened on appropriately.

Low-frequency ultrasound is used to image the abdominal cavity and pericardium in these patients, using either a curvilinear transducer or a phased-array transducer. Both of these transducers are capable of acquiring the images necessary to interpret a FAST exam, but it has not been well studied whether using one transducer instead of the other improves time to image acquisition or image quality.

In this study, physician ultrasound operators are asked to perform FAST exams on healthy non-injured volunteers for the purpose of determining if there is a difference in the time to acquisition or quality of images between phased-array and curvilinear transducers.

ELIGIBILITY:
Inclusion Criteria:

Study's ultrasound operators must be emergency medicine residents or PA/NP fellows currently enrolled in an emergency medicine training program between the ages of 18 - 64 years who are not pregnant.

Study's healthy normal volunteers must be emergency medicine faculty, fellows, or PA/NPs aged 18-64 with no anatomic abnormalities, prior surgeries, or significant chronic medical conditions.

Exclusion Criteria:

Pregnant women

Prisoners

Anyone below the age of 18 or above the age of 64 years old

Individuals with abnormal/thoracic anatomy (such as individuals with situs inversus) and individuals with chronic medical conditions that would limit their ability to participate in the study or have ultrasound images taken of them.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-27 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Time Required | Assessed and reported at study completion, estimated 1 year
  Total time necessary to perform a FAST ultrasound examination using either transducer specified, starting from when the exam is begun to when the last view is completed by the ultrasound operator. The average exam is estimated to take no more than 10 minutes to complete.

SECONDARY OUTCOMES:
Image Quality | Assessed and reported at study completion, estimated 1 year
  Quality of the images, based on retrospectively reviewing and assessing the interpretability of sonographic images taken during the FAST exam performed with either transducer. These images are captured during the performance of the ultrasound exam.

CONTACTS AND LOCATIONS:
Overall Officials: Sherwin A Soltani, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.

DOCUMENTS (2):
  • Study Protocol (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT04333680/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT04333680/SAP_001.pdf